CLINICAL TRIAL: NCT01676532
Title: Feasibility Study on the Model School Pediatric Health Initiative Pilot Project
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jonathon Maguire, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000025631
Record Dates: First submitted 2012-08-21; First posted 2012-08-31 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: School Board Health Centers
Keywords: School Board Health Center; Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Students attending SBHC: Students who attend the SBHC from either Sprucecourt Public School or any other participating schools.
  Interventions: Other: Students attending SBHC

INTERVENTIONS:
Other: Students attending SBHC — School based health clinic. This is a cohort study as such there is only one group of children who used the SBHC

SUMMARY:
This is a prospective cross sectional study to assess the feasibility of a school based health centre (SBHC) at Sprucecourt Public School, an inner-city elementary school in Toronto. The SBHC allows inner-city children who face barriers to accessing health care the opportunity to receive health care in their school.The primary aim of this study is to determine utilization of the SBHC. Establishing feasibility of the SBHC would support further development and expansion of this program into other inner city schools.

DETAILED DESCRIPTION:
A chart review of the first year of the SBHC was conducted. Feasibility metrics included the number of children who enrolled at the SBHC. Efficacy metrics included the proportion of enrolled children who enrolled at SBHC. Efficacy metrics included the proportion of enrolled children who attended and received new diagnoses and treatment plans

ELIGIBILITY:
Inclusion Criteria:

* All students at Sprucecourt Public School and the surrounding fourteen schools, as well as their siblings (ages 0-12 years), who are enrolled at and have consent to attend the SBHC
* All infants and preschool aged children attending the on-site Parenting and Family Literacy Centre who are enrolled at the SBHC

Exclusion Criteria:

* N/A

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All students of Sprucecourt Public School as well as the fourteen surrounding inner city public schools and their siblings. All children attending the on-site Parenting and Family Literacy Centre.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Maguire, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Students Attending SBHC
Started | 127
Completed | 127
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Students Attending SBHC
Number analyzed (Participants) | 127
Age, Categorical [Count of Participants; unit: Participants] — Retrospective chart review
  Participants
    <=18 years | 127
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 127
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 95
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 10
  More than one race | 8
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Enrolled Participants Who Attended SBHC
Description: The primary objectives are to determine utilization of the SBHC including:
  1. The number of students who are enrolled at the SBHC
  2. The number of enrolled students enrolled who attended the SBHC
Time Frame: 1 year
Population: 379 students enrolled in the SBHC and 127 of those students attended SBHC. Existing data is based on 127 students who attended SBHC.
Measure: Number; unit: participants
Groups:
- Students Attending SBHC: Students who were enrolled at the SBHC and then attended the SBHC
Arm/Group | Students Attending SBHC
Number analyzed (Participants) | 379
participants
  Total number of students attending SBHC | 127
  Number of students not attending SBHC | 252

2. Secondary Outcome: Number of Students Attending SBHC With New Treatment Plans
Description: Proportion of children seen in the clinic with treatment plans
Time Frame: 1 year
Population: 115 students out of 127 students attending SBHC had a new treatment plan.
Measure: Number; unit: participants
Groups:
- Number of Students Attending SBHC With New Treatment Plans: The total number of students who attended SBHC that had new treatment plans proposed
Arm/Group | Number of Students Attending SBHC With New Treatment Plans
Number analyzed (Participants) | 127
participants
  Number of students with treatment plans | 115
  Number of students with no treatment plans | 12

3. Secondary Outcome: Number of Students Attending SBHC With New Diagnoses
Description: Number of students attending SBHC with new diagnoses
Time Frame: 1 year
Population: 120 of the 127 students who attended the SBHC had a new diagnosis. 94 received one new diagnosis and 26 children received more than one new diagnosis
Measure: Number; unit: participants
Groups:
- Number of Students Attending SBHC With New Diagnoses: Porportion of students attending SBHC with new diagnoses
Arm/Group | Number of Students Attending SBHC With New Diagnoses
Number analyzed (Participants) | 127
participants
  Number of students attending SBHC_ new diagnosis | 94
  Number of students attending SBHC with >1 new diag | 26
  No new diagnosis | 7

4. Secondary Outcome: Number of Referrals Made of Students Attending SBHC
Description: Number of referrals of the 127 students who attended the SBHC from 8 months-1 year of the opening of the clinic
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Number of Referrals Made for Students Attending SBHC: Types and number of referrals made for students attending SBHC.
Arm/Group | Number of Referrals Made for Students Attending SBHC
Number analyzed (Participants) | 127
participants
  Number of students with no referrals | 97
  number of students referred to family physician | 20
  number of students referred to specialist | 10
  number of students referred for psychological test | 6
  number of students ref to community mental health | 3
  number of students referred to dietician | 1
  number of students referred to audiology testing | 19
  number of students referred to vision testing | 7

5. Other Pre Specified Outcome: Number of Students Enrolled in SBHC Who Were From the Host School (Sprucecourt)
Description: The number of students who enrolled in SBHC who were from the host school Sprucecourt
Time Frame: 8 months
Population: Total number of students who enrolled in SBHC. Outcome is the number of students from host school (sprucecourt) who enrolled in SBHC
Measure: Number; unit: participants
Groups:
- Number of Students From Sprucecourt Who Enrolled in SBHC: From the total number of students who enrolled in the SBHC, the number of students from the host school (Sprucecourt) was calculated
Arm/Group | Number of Students From Sprucecourt Who Enrolled in SBHC
Number analyzed (Participants) | 379
participants | 227

6. Other Pre Specified Outcome: Sprucecourt Public School Vs Other Participating Schools
Description: To compare the number of students who attend the SBHC from the host school (Sprucecourt Public School) with the number of students who attend the SBHC from the other participating schools
Time Frame: 8 months
Population: total number of students who attended SBHC
Measure: Number; unit: participants
Groups:
- Sprucecourt Public School Vs Other Participating Schools: The number of students from the host school of the SBHC and other participating schools
Arm/Group | Sprucecourt Public School Vs Other Participating Schools
Number analyzed (Participants) | 127
participants
  number of students attending from Sprucecourt | 89
  number of students attending from school cluster | 20
  number of students attending from preschool age | 14
  number of students with unknown enrolment data | 4

7. Other Pre Specified Outcome: Number of Students Triaged From School Support Team Meetings
Description: The number of students triaged from SST meetings was not collected.
Time Frame: 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Students Referred to SBHC Who Attended SBHC
Description: This data was not collected.
Time Frame: 8 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Follow-up Appointments
Description: Attendance at follow-up appoints was not collected.
Time Frame: 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Absenteeism
Description: Outcome data comparing absenteeism in the school with the year preceding the SBHC was not collected
Time Frame: 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Ontario Health Insurance Plan (OHIP)Status
Description: OHIP status of students attending the clinic was not reported or collected
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: no adverse events were reported for students attending SBHC
Arm/Group | Students Attending SBHC
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No